CLINICAL TRIAL: NCT06524752
Title: Risk Factors for Postoperative Nausea and Vomiting in Patients Undergoing Day-case Hysteroscopic Surgery
Brief Title: Risk Factors for PONV in Patients Undergoing Hysteroscopic Surgery
Status: Completed | Type: Observational
Sponsor: Weifang Medical University (Other)
Responsible Party: Principal Investigator, Jiang Liu, Research investigator, Weifang Medical University
Other Study IDs: KYLL20230217-3
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Gynecologic Nursing; Postoperative Complications
Keywords: PONV; Risk factor; Nursing
MeSH Terms: conditions — Postoperative Complications; Postoperative Nausea and Vomiting | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: The patient experience the postoperative nausea or vomiting
  Interventions: Other: The presence of nausea and vomiting within 24 hours after surgery
- Control group: The patient did not experience postoperative nausea or vomiting
  Interventions: Other: Non-existence of nausea and vomiting within 24 hours after surgery

INTERVENTIONS:
Other: The presence of nausea and vomiting within 24 hours after surgery — This is a prospective risk prediction model building, thus there is no traditional definition of intervention.
  Groups: Observation group
Other: Non-existence of nausea and vomiting within 24 hours after surgery — This is a prospective risk prediction model building, thus there is no traditional definition of intervention.
  Groups: Control group

SUMMARY:
The purpose of this study was to construct and validate a risk prediction model for PONV in patients undergoing hysteroscopic day-case surgery.

DETAILED DESCRIPTION:
This study predicted the risk of postoperative nausea and vomiting in patients undergoing day-case hysteroscopic surgery by constructing and validating a web-based dynamic nomogram.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing hysteroscopic day-case surgery and aged 18 years.

Exclusion Criteria:

* Patients with intraoperative change of surgical method and unstable postoperative vital signs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The objective of this study was to develop a risk prediction model for postoperative nausea and vomiting in patients undergoing day-case hysteroscopic surgery. Therefore, the target population of this study was limited to female patients with gynecologic diseases and requiring day-case hysteroscopic surgery.
Study Population: Female patients undergoing gynaecological hysteroscopic day-case surgery.
Sampling Method: Probability Sample
Enrollment: 1583 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
PONV | Within 24 hours after surgery
  The occurrence and severity of PONV is evaluated by Visual Analogue Scale (VAS). The VAS scale ranges from 0 to 10, with larger scores meaning that the patient has more severe PONV.

CONTACTS AND LOCATIONS:
Overall Officials: Shirong Fang, Researcher, Study Director — Weifang People's Hospital
Locations (1):
- Weifang People's Hospital, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No